CLINICAL TRIAL: NCT06574763
Title: Neoadjuvant RC48 Plus Carboplatin for HER2-expressing Advanced Ovarian Cancer: a Prospective Phase 2 Exploratory Study
Brief Title: Neoadjuvant RC48 Plus Carboplatin for HER2-expressing Advanced Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jundong Li, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-318-01
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48+Carboplatin (Experimental)
  Interventions: Drug: RC48/Carboplatin

INTERVENTIONS:
Drug: RC48/Carboplatin — RC48, 2.5mg/kg, iv, Q3W Carboplatin, AUC 5, iv, D1, Q3W

SUMMARY:
The goal of this phase II single arm prospective clinical study is to evaluate the efficacy and toxicity of RC48 plus carboplatin neoadjuvant therapy in HER2 expressed epithelial ovarian cancer patients. The main questions it aims to answer are:

* The improvement of complete resection rate and pathological complete rate of this regimen.
* The delayed effect of treatment regimens on patient's recurrence.

DETAILED DESCRIPTION:
The current standard treatment for newly diagnosed ovarian cancer involves a combination of surgery, chemotherapy, and adjuvant therapy. Ovarian cancer surgery is challenging and has a high incidence of postoperative complications. Many studies have explored the use of neoadjuvant therapy before surgery to shrink tumors and downstage the disease, aiming to increase the proportion of operable patients and the rate of complete resection, while also reducing surgical difficulty and associated risks. Guidelines recommend that neoadjuvant chemotherapy for high-grade serous ovarian cancer should be consistent with the first-line chemotherapy regimen, with paclitaxel/carboplatin every three weeks being the preferred regimen in clinical practice.

However, there are still unmet needs in neoadjuvant chemotherapy for ovarian cancer: 1. The rate of pathologic complete response (pCR) after neoadjuvant chemotherapy is less than 10%, yet achieving pCR significantly improves prognosis; 2. Using the same regimen for neoadjuvant chemotherapy and postoperative chemotherapy may lead to the development of subsequent chemotherapy resistance, thereby shortening the time before the patient develops platinum resistance; 3. Neoadjuvant chemotherapy can have severe adverse reactions.

RC48 (Disitamab Vedotin) is a human epidermal growth factor 2 (HER2)-directed antibody-drug conjugate, with a novel humanized anti-HER2 antibody disitamab conjugated to monomethyl auristatin E (MMAE) via a cleavable linker. This study used RC48 combined with carboplatin to explore the efficacy and toxic side effects of this regimen as neoadjuvant therapy in epithelial ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

- General criteria:

1. Voluntarily consent to participate in the study and sign an informed consent form.
2. Age 18-75 years (at the time of signing consent).
3. Expected survival ≥ 12 months.
4. ECOG performance status 0 or 1.
5. Body weight must be >30 kg.
6. Able to understand trial requirements and willing and able to adhere to trial and follow-up procedures.
7. Women of childbearing potential (defined as not having undergone surgical sterilization or not having naturally menstruated for at least 12 consecutive months) must agree to use effective contraception during the study treatment.

   - Tumor-related criteria:
8. Newly diagnosed, histologically or cytologically confirmed FIGO stage III-IV high-grade serous ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
9. HER2 expression: including patients with HER2 immunohistochemistry (IHC) results of IHC 1+ or higher and gene amplification detected by ERBB2 testing.
10. Physical condition unsuitable for direct surgery or imaging or laparoscopic assessment indicating low likelihood of achieving complete resection through direct surgery.
11. Patients must have at least one measurable lesion according to RECIST v1.1 criteria (assessed by the investigator).

    - Adequate organ function: Criteria met within 28 days prior to the first dose of Cycle 1:
12. Bone marrow function:

    Hemoglobin ≥ 90 g/dL Absolute neutrophil count ≥ 1.5 × 10^9/L Platelet count ≥ 100 × 10^9/L
13. Liver function (normal values as defined by the clinical trial center):

    Serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN) In the absence of liver metastases, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 2.5 × ULN; with liver metastases, ALT, AST, and ALP ≤ 5 × ULN
14. Renal function (normal values as defined by the clinical trial center):

    Serum creatinine ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 50 mL/min (Cockcroft-Gault formula) Urinalysis showing urinary protein ≥ 3+ should be followed by a 24-hour urine collection with 24-hour urinary protein < 3.5 g
15. Coagulation function:

    International normalized ratio (INR) ≤ 1.5 or 2.5 (for patients receiving anticoagulation therapy) Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN
16. Cardiac function:

New York Heart Association (NYHA) classification < Grade 3

Exclusion Criteria:

- Tumor-related criteria:

1. Histologic types of endometrioid carcinoma, clear cell carcinoma, mucinous carcinoma, or sarcomatoid tumors, including any mixed tumors with these types, or low-grade/borderline ovarian tumors.
2. Known active central nervous system (CNS) metastases and/or leptomeningeal disease.
3. Presence of pleural effusion, pericardial effusion, or ascites that cannot be controlled through drainage or other methods.

   - Comorbidities and medical history:
4. Severe clinically significant active infections.
5. History of multiple sclerosis (MS) or other demyelinating diseases and/or Lambert-Eaton syndrome (paraneoplastic syndrome).
6. Significant clinically relevant heart disease, including but not limited to:

   1. Myocardial infarction within ≤ 6 months prior to first dose;
   2. Unstable angina;
   3. Uncontrolled congestive heart failure (> II grade);
   4. Uncontrolled hypertension (≥ 3 grade per CTCAE criteria);
   5. Uncontrolled arrhythmias.
7. Cerebrovascular accident (CVA), transient ischemic attack (TIA), or intracranial hemorrhage (e.g., brain hemorrhage, subarachnoid hemorrhage, or subdural hemorrhage) within 6 months prior to enrollment.
8. ECG showing clinically significant abnormal results.
9. History of clinically diagnosed and currently active non-infectious interstitial lung disease (ILD), including non-infectious pneumonia, pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-induced pneumonitis, or other severe pulmonary diseases.
10. History of liver cirrhosis (Child-Pugh class C).
11. History of abdominal wall fistula, gastrointestinal perforation, or active gastrointestinal bleeding within 6 months prior to randomization.
12. Bleeding disorders or significant coagulation abnormalities (in the absence of anticoagulation).
13. Major surgery within 4 weeks prior to enrollment (except for exploratory procedures performed at other institutions).
14. Non-healing wounds, active ulcers, or fractures.
15. History of other primary malignancies, except for those with minimal risk of metastasis or death.

    - Concurrent treatments:
16. Previous treatment with Vedicimab or other HER2-targeted therapies.
17. Prior anti-cancer treatment for ovarian cancer, including chemotherapy, immunotherapy, or targeted therapy; patients may receive concurrent hormone therapy (e.g., hormone replacement therapy) or bisphosphonates for non-cancer-related conditions.

    - Other:
18. Known hypersensitivity to monoclonal antibody therapy, MMAE class drugs, or any component of the study drug.
19. Pregnant or breastfeeding women.
20. Investigator believes the subject has other severe systemic diseases or conditions that make participation in the clinical study inappropriate.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Completed Resection Rate | 3-month
  Completed Resection Rate (CRR): Complete tumor resection is defined as the absence of gross residual intra-abdominal and pelvic lesions assessed by the investigator during interval debulking surgery after the patient has received neoadjuvant therapy. The CRR is the percentage of patients achieving complete tumor resection.

SECONDARY OUTCOMES:
Pathologic complete response | 3-month
  percentage of patients who achieved complete response
Objective Response Rate (ORR) | 3-month
  Objective tumor response was defined as the proportion of patients whose tumor volume has been reduced to a predetermined value and can be maintained for more than 3 cycles, ie ORR=CR+PR
Progression Free Survival (PFS) | 3-year
  Progression-free survival was defined as the duration of time from study entry to time of progression, death, or the date of last contact, whichever occurs first
Adverse Event Rate | from the first day of treatment till 30 days after discontinuing the medication
  The Adverse Event Rate is defined as the percentage of patients who experience any Adverse Events (AE), Serious Adverse Events (sAE), and Treatment-Related Adverse Events (TEAEs) from the first day of treatment till 2 years after discontinuing the medication
Overall survival | 5-year
  OS is defined as the time from the study enrollment to death due to any cause.